CLINICAL TRIAL: NCT06527482
Title: A Multicenter Prospective Cohort Study of Autologous Osteoperiosteal Transplantation for the Treatment of Severe Osteochondral Lesions of the Talus
Brief Title: Autologous Osteoperiosteal Transplantation for the Treatment of Severe Osteochondral Lesions of the Talus
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2023418
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-06

CONDITIONS: Osteochondral Lesion of Talus; Autologous Osteoperiosteal Transplantation
Keywords: Osteochondral Lesion of Talus; Autologous Osteoperiosteal Transplantation; Arthroscopic Techniques; Clinical Efficacy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Autologous Osteoperiosteal Transplantation — After full exposure of the lesion, the center of the cystic lesion was determined and drilled perpendicularly using a 2-mm pin. Then, a 4.5-mm cannulated bore was used to drill the lesion until the cyst was reached, and a small bone socket was created. A harvester tube matching the diameter of the cyst was used to enlarge the bone socket with care to avoid damage to the adjacent normal cartilage. The cystic lesion was debrided thoroughly, and the sclerotic wall of the cyst was freshened using a curette. The harvester tube with a matched diameter was driven in to a depth of 15 to 20 mm at the 2-cm proximal part of the anterior superior iliac spine perpendicularly without violation of the lateral wall of the crest. When necessary, small pieces of cancellous bone were also harvested from the iliac crest using a bone curette then grafted into the peripheral area of the cyst to fill up the remaining space of the cyst around the bone socket in the talus.

SUMMARY:
The goal of this clinical trial is to establish a multicenter prospective cohort of patients with severe osteochondral lesion of the talus (OLT), evaluate the clinical efficacy of autologous osteoperiosteal transplantation and the incidence of postoperative donor-site morbidity. The main questions it aims to answer are:

Does autologous osteoperiosteal transplantation have good clinical outcomes in the treatment of severe OLT? Does autologous osteoperiosteal transplantation treat severe OLT with fewer postoperative complications?

Participants will:

Undergo autologous osteoperiosteal transplantation for OLT Receive clinical follow-up 3, 6, 12, and 24 months after surgery and answer scales of ankle function assessment Take CT and MRI preoperatively and 12 and 24 months after surgery

ELIGIBILITY:
Inclusion Criteria:

* Chronic ankle pain, diagnosed as Osteochondral Lesions of the Talus (OLT);
* Hepple V OLT on the medial side of the talus or the diameter of the lesion ≥ 8 mm;
* Conservative treatment of at least 3 months fails to relieve symptoms;
* Willingness to voluntarily participate in the trial and to sign informed consent.

Exclusion Criteria:

* Varus or valgus deformity of the ankle of more than 5 degrees;
* Grade III injury of the lateral collateral ligament of ankle;
* Chronic synovitis (rheumatoid arthritis, pigmented villous nodular synovitis, etc.);
* Joint fibrosis, stiffness, and significantly restricted range of motion;
* Evidence of moderate to severe knee osteoarthritis on plain radiographs;
* Failure to complete the rehabilitation protocol as required;
* Patient medically not fit for surgery, radiographs or MRI;
* For women, pregnant, planning to be pregnant or lactating.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Severe OLT patients undergoing autologous osteoperiosteal transplantation that meet the above criteria
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Foot and Ankle Outcome Score (FAOS) | Pre-surgery and 6 weeks and 3, 6, 12 and 24 months after surgery
  The Foot and Ankle Outcome Score (FAOS) is an extensive tool designed to evaluate the patient's perception of their foot and ankle conditions, with 0 indicating the worst possible outcome, and 100 representing the best possible outcome. The scale of FAOS score will be answered by participants during clinic follow-up preoperatively, and 6 weeks 3, 6, 12 and 24 months after surgery.

SECONDARY OUTCOMES:
American Orthopedic Foot and Ankle Society Score (AOFAS) | Pre-surgery and 6 weeks and 3, 6, 12 and 24 months after surgery
  The AOFAS is a standardized tool used to evaluate the outcomes of treatments for foot and ankle disorders, with 0 indicating severe disability or extreme problems, and 100 indicating no disability or problems.The scale of AOFAS score will be answered by participants during clinic follow-up preoperatively, and 6 weeks 3, 6, 12 and 24 months after surgery.
Visual Analogue Scale (VAS) | Pre-surgery and 6 weeks and 3, 6, 12 and 24 months after surgery
  The Visual Analog Scale (VAS) is a simple and widely used method for assessing the intensity of pain and other subjective experiences, with 0 indicating no pain, and 100 indicating the worst possible pain. The scale of VAS score will be answered by participants during clinic follow-up preoperatively, and 6 weeks 3, 6, 12 and 24 months after surgery.
Ankle Activity Score (AAS) | Pre-surgery and 6 weeks and 3, 6, 12 and 24 months after surgery
  The AAS is a scoring tool to assess sports activity for the ankle joint, with zero point indicating the lowest activity level, and ten points indicating the highest activity level. The scale of AAS score will be answered by participants during clinic follow-up preoperatively, and 6 weeks 3, 6, 12 and 24 months after surgery.
Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) | 12 and 24 months after surgery
  The Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) score is a grading system used to evaluate the quality of cartilage repair tissue through MRI (Magnetic Resonance Imaging), with 0 indicating poor cartilage repair quality, and 100 indicating excellent cartilage repair quality. MOCART score will be assessed on magnetic resonance imaging 12 and 24 months after surgery.
International Cartilage Repair Society (ICRS) | 12 months after surgery
  The International Cartilage Repair Society (ICRS) score is a grading system used to assess the condition of articular cartilage, especially in the context of cartilage repair procedures, with 0 indicating poor cartilage repair quality, and 12 indicating excellent cartilage repair quality. ICRS score will be assessed 12 months
Complications | Final follow-up (48 months after surgery)
  Complications, including infection,hematoma, stiffness, recurrent ankle pain will be continuously followed during clinic follow-up and will be overall collected 24 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Qinwei Guo, MD, Principal Investigator — Department of Sports Medicine, Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China